CLINICAL TRIAL: NCT01037322
Title: Use of Cannabidiol for the Treatment of Inflammatory Bowel Disease
Brief Title: Cannabidiol for Inflammatory Bowel Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, NAFTALI TIMNA, MD, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: canabidiol1
Record Dates: First submitted 2009-12-20; First posted 2009-12-23 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: crohn's disease; ulcerative colitis; cannabis; cannabidiol
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Marijuana Abuse | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- cannabidiol in drops (Active Comparator): cannabidiol given in drops of olive oil sub lingual 5 mg twice daily
  Interventions: Drug: cannabidiol
- placebo in drops (Placebo Comparator): olive oil given in drops sub lingual
  Interventions: Drug: placebo in drops

INTERVENTIONS:
Drug: cannabidiol — cannabidiol given in olive oil drops, 5 mg twice daily
  Arms: cannabidiol in drops
Drug: placebo in drops — olive oil containing no drug given in drops twice daily
  Arms: placebo in drops

SUMMARY:
There are many anecdotal reports about improvement of Inflammatory bowel diseases (IBD) with cannabis smoking. The most effective anti inflammatory compound known today is cannabidiol. cannabidiol can be extracted from the cannabis plant, it has no central effect and is fat soluble so it can be given as drops in oil. Doses of up to 500mg did not cause any side effects.

The aim of the proposed study is to examine in a double blind placebo controlled fashion the effect of cannabidiol on disease activity in patients with IBD.

DETAILED DESCRIPTION:
Background: Inflammatory bowel diseases (IBD) are relatively common disease with a rising incidence. Treatment includes various immunocompromising agents including corticosteroids, immunomodulators and biologic agents. Current treatment is not always effective and has many side effect.

Cannabinoids have been known to have anti inflammatory effect, probably via the CB2 receptor. There are many anecdotal reports of cannabinoids in inflammatory disease such as rheumatoid arthritis, and the impression is that cannabinoids do have an ameliorating effect on IBD and that side effects are negligible. However, there are no placebo controled trials in human subjects.

The cannabis plant contains about 600 ingredients, and it is not known which are the active ingredients affecting IBD. The most effective anti inflammatory compound known today is cannabidiol. Cannabidiol can be extracted from the cannabis plant, it has no central effect and is fat soluble so it can be given as drops in oil. Doses of up to 500mg did not cause any side effects.

The aim of the proposed study is to examine in a double blind placebo controlled fashion the effect of cannabidiol on disease activity in patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis IBD at least 3 months before recruitment will be eligible to the study.
2. Patients with active disease who are resistant to either 5 ASA, steroids or immunomodulators, or who can not receive those drugs due to adverse reactions will be offered the possibility of receiving cannabidiol at a dose of 10 mg in sub lingual drops or drops of olive oil as placebo.
3. Disease activity index of either CDAI of more then 200 in Crohn's disease or Mayo score above 3 in UC.
4. Age above 20.

Exclusion Criteria:

1. Patients with a known mental disorder
2. Patients who are deemed to be at a high risk of abuse or addiction to the study drug.
3. Pregnant women
4. Patients who are sensitive to any of the ingredients of the study medication.
5. Patients who are unable to give informed consent.
6. Patients who may need surgery in the near future.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
reduction of 70 points in CDAI | 8 weeks

SECONDARY OUTCOMES:
change in quality of life during the study | 8 weeks
any adverse events during study period | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fred Konikoff, professor, Study Chair — Meir Hospital
Locations (1):
- Sapir Medical center Meir Hospital, Kfar Saba, Israel

REFERENCES:
- [Derived] Naftali T, Mechulam R, Marii A, Gabay G, Stein A, Bronshtain M, Laish I, Benjaminov F, Konikoff FM. Low-Dose Cannabidiol Is Safe but Not Effective in the Treatment for Crohn's Disease, a Randomized Controlled Trial. Dig Dis Sci. 2017 Jun;62(6):1615-1620. doi: 10.1007/s10620-017-4540-z. Epub 2017 Mar 27. PMID 28349233